CLINICAL TRIAL: NCT02270008
Title: Reducing Perinatal Anal Incontinence Through Early Pelvic Floor Muscle Training: a Prospective Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Deborah Karp, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00065572
Record Dates: First submitted 2014-07-14; First posted 2014-10-21 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Perinatal and Postpartum Anal Incontinence
Keywords: anal incontinence; pregnancy-associated pelvic floor disorders
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pelvic floor training (Active Comparator): The intervention group will undergo an in-person standardized training session by a trained nurse practitioner. The intervention is the pelvic floor training session. They will then be asked to continue muscle training at home at regular intervals and asked to log their exercises on a standardized exercise diary that is provided to them.
  Interventions: Other: Pelvic floor training
- Literature-only group (No Intervention): The literature-only group will receive a pamphlet with instructions for pelvic floor muscle exercises; however, no in-person training will be administered.

INTERVENTIONS:
Other: Pelvic floor training — Baseline muscle strength will be measured with the modified Oxford scale. The intervention group will undergo an in-person standardized pelvic strength training session by a trained nurse practitioner.
  Arms: Pelvic floor training

SUMMARY:
Anal incontinence affects up to 20% of gravid women during and immediately after pregnancy. It can lead to embarrassment, poor self-image, lifestyle changes, in addition to poor hygiene and increased risk for genitourinary tract infection. These women suffer from a combination of loss of fecal and/or flatal control, with increasing frequency as pregnancy progresses. Though anal incontinence may subside in the postpartum period, a subset of women will have continued anal incontinence or recurrence of anal incontinence with subsequent pregnancies or as they age. As of December 2012, only one study has explored the effects of pelvic floor muscle training (PFMT) on reducing the development of this condition in the pregnant population. However, that study took place in Scandinavia with little demographic correlation to a US population and lacked postpartum followup. Although their results showed little effect of PFMT on anal incontinence, they recommended further research to be performed prior to making definitive conclusions.

Multiple studies have explored the effects of PFMT on urinary incontinence, and the general consensus shows a positive benefit, with a 50% incidence reduction. This study will serve as an initial test to explore whether such a positive relationship holds for anal incontinence throughout pregnancy and postpartum period for a diverse population. The format will be a prospective feasibility trial comprised of a one-time intensive in-person pelvic floor muscle training course at the first prenatal visit with at home instructions for continued exercise. This group will be compared to a control group which receives a hand-out regarding PFMT but no personalized instruction. The progress of the participants and their symptoms of incontinence will be monitored during pregnancy and at the postpartum visit using standardized validated pelvic floor questionnaires, based on previously designed surveys. A sample size of 100 parous women ages 20-35 year old will be randomized to an intervention and "control or standard therapy" group. The investigators' hypothesis is that the intervention group will show a 50% risk reduction, similar to the urinary incontinence studies. The results of this study will then allow us to design a broader intervention study for which to study the effects of PFMT and anal incontinence during pregnancy and the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* parous women
* ages 20-40year old
* a new Ob visit prior to 20 weeks gestation
* confirmed singleton live intrauterine pregnancy

Exclusion Criteria:

* prior history of anal incontinence or prolapse
* history of surgery or procedures for urinary or anal incontinence or pelvic organ prolapse
* tobacco use
* diabetes mellitus
* history of sexual trauma
* chronic cough
* chronic constipation based on Rome criteria
* known connective tissue disorder

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence of fecal and/or flatal incontinence | 3 months (1st trimester)
  based on standardized questionnaires
Incidence of fecal and/or flatal incontinence | 6 months (2nd trimester)
  based on standardized questionnaires
Incidence of fecal and/or flatal incontinence | 9 months (3rd trimester)
  based on standardized questionnaires

SECONDARY OUTCOMES:
Exercise compliance | 3 months (1st trimester)
  patient-reported pelvic floor exercise diary
Exercise compliance | 6 months (2nd trimester)
  patient-reported pelvic floor exercise diary
Exercise compliance | 9 months (3rd trimester)
  patient-reported pelvic floor exercise diary

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Karp, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Department of Obstetrics and Gynecology Clinic, Atlanta, Georgia, United States

REFERENCES:
- [Background] Bo K, A H Haakstad L, Voldner N. Do pregnant women exercise their pelvic floor muscles? Int Urogynecol J Pelvic Floor Dysfunct. 2007 Jul;18(7):733-6. doi: 10.1007/s00192-006-0235-2. Epub 2006 Nov 21. PMID 17120174
- [Background] Brown SJ, Donath S, MacArthur C, McDonald EA, Krastev AH. Urinary incontinence in nulliparous women before and during pregnancy: prevalence, incidence, and associated risk factors. Int Urogynecol J. 2010 Feb;21(2):193-202. doi: 10.1007/s00192-009-1011-x. Epub 2009 Oct 16. PMID 19834637
- [Background] Eason E, Labrecque M, Marcoux S, Mondor M. Anal incontinence after childbirth. CMAJ. 2002 Feb 5;166(3):326-30. PMID 11868640
- [Background] Fine P, Burgio K, Borello-France D, Richter H, Whitehead W, Weber A, Brown M; Pelvic Floor Disorders Network. Teaching and practicing of pelvic floor muscle exercises in primiparous women during pregnancy and the postpartum period. Am J Obstet Gynecol. 2007 Jul;197(1):107.e1-5. doi: 10.1016/j.ajog.2007.02.052. PMID 17618779
- [Background] Fynes MM, Marshall K, Cassidy M, Behan M, Walsh D, O'Connell PR, O'Herlihy C. A prospective, randomized study comparing the effect of augmented biofeedback with sensory biofeedback alone on fecal incontinence after obstetric trauma. Dis Colon Rectum. 1999 Jun;42(6):753-8; discussion 758-61. doi: 10.1007/BF02236930. PMID 10378599
- [Background] Glazener CM, Herbison GP, MacArthur C, Grant A, Wilson PD. Randomised controlled trial of conservative management of postnatal urinary and faecal incontinence: six year follow up. BMJ. 2005 Feb 12;330(7487):337. doi: 10.1136/bmj.38320.613461.82. Epub 2004 Dec 22. PMID 15615766
- [Background] Glazener CM, Herbison GP, Wilson PD, MacArthur C, Lang GD, Gee H, Grant AM. Conservative management of persistent postnatal urinary and faecal incontinence: randomised controlled trial. BMJ. 2001 Sep 15;323(7313):593-6. doi: 10.1136/bmj.323.7313.593. PMID 11557703
- [Background] Hay-Smith J, Morkved S, Fairbrother KA, Herbison GP. Pelvic floor muscle training for prevention and treatment of urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD007471. doi: 10.1002/14651858.CD007471. PMID 18843750
- [Background] MacArthur C, Wilson D, Herbison P, Lancashire RJ, Hagen S, Toozs-Hobson P, Dean N, Glazener C; ProLong study group. Faecal incontinence persisting after childbirth: a 12 year longitudinal study. BJOG. 2013 Jan;120(2):169-179. doi: 10.1111/1471-0528.12039. Epub 2012 Nov 27. PMID 23190303
- [Background] Morkved S, Bo K, Schei B, Salvesen KA. Pelvic floor muscle training during pregnancy to prevent urinary incontinence: a single-blind randomized controlled trial. Obstet Gynecol. 2003 Feb;101(2):313-9. doi: 10.1016/s0029-7844(02)02711-4. PMID 12576255
- [Background] Pollack J, Nordenstam J, Brismar S, Lopez A, Altman D, Zetterstrom J. Anal incontinence after vaginal delivery: a five-year prospective cohort study. Obstet Gynecol. 2004 Dec;104(6):1397-402. doi: 10.1097/01.AOG.0000147597.45349.e8. PMID 15572505
- [Background] Reilly ET, Freeman RM, Waterfield MR, Waterfield AE, Steggles P, Pedlar F. Prevention of postpartum stress incontinence in primigravidae with increased bladder neck mobility: a randomised controlled trial of antenatal pelvic floor exercises. BJOG. 2002 Jan;109(1):68-76. doi: 10.1111/j.1471-0528.2002.t01-1-01116.x. PMID 11845813
- [Background] Rortveit G, Daltveit AK, Hannestad YS, Hunskaar S; Norwegian EPINCONT Study. Urinary incontinence after vaginal delivery or cesarean section. N Engl J Med. 2003 Mar 6;348(10):900-7. doi: 10.1056/NEJMoa021788. PMID 12621134
- [Background] Signorello LB, Harlow BL, Chekos AK, Repke JT. Midline episiotomy and anal incontinence: retrospective cohort study. BMJ. 2000 Jan 8;320(7227):86-90. doi: 10.1136/bmj.320.7227.86. PMID 10625261
- [Background] Stafne SN, Salvesen KA, Romundstad PR, Torjusen IH, Morkved S. Does regular exercise including pelvic floor muscle training prevent urinary and anal incontinence during pregnancy? A randomised controlled trial. BJOG. 2012 Sep;119(10):1270-80. doi: 10.1111/j.1471-0528.2012.03426.x. Epub 2012 Jul 17. PMID 22804796
- [Background] Wesnes SL, Rortveit G, Bo K, Hunskaar S. Urinary incontinence during pregnancy. Obstet Gynecol. 2007 Apr;109(4):922-8. doi: 10.1097/01.AOG.0000257120.23260.00. PMID 17400855
- [Background] Whitford HM, Jones M. An exploration of the motivation of pregnant women to perform pelvic floor exercises using the revised theory of planned behaviour. Br J Health Psychol. 2011 Nov;16(4):761-78. doi: 10.1111/j.2044-8287.2010.02013.x. Epub 2011 Jan 13. PMID 21988063
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735